CLINICAL TRIAL: NCT03095599
Title: A Phase 2/3 Double Blinded, Randomized, Placebo-Controlled Study in Healthy Adult Volunteers in Vietnam to Examine the Safety and Immunogenicity of a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine (IVACFLU-S) Produced by IVAC
Brief Title: Seasonal Trivalent Inactivated Split Virion Influenza Vaccine Clinical Trial (IVACFLU-S) - PHASE 2/3
Acronym: IVACFLUS-0203
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Vaccines and Medical Biologicals, Vietnam (Industry)
Collaborators: Pasteur Institute, Ho Chi Minh City (Other Government); PATH (Other); Quintiles, Inc. (Industry); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IVACFLU-S 0203; CVIA 051 (Other: PATH)
Record Dates: First submitted 2017-03-13; First posted 2017-03-29 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Influenza, Human
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): Received one dose of IVACFLU-S vaccine intramuscularly.
  Interventions: Biological: IVACFLU-S
- Placebo (Placebo Comparator): Received one dose of placebo intramuscularly.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IVACFLU-S — IVACFLU-S is seasonal inactivated, split virion, trivalent influenza vaccine (A/H3N2, A/H1N1, and B), produced in GCP facility by IVAC uses embryonated chicken eggs. This vaccine is purified by sucrose gradient ultracentrifugation (Alfa Wassermann, West Caldwell, NJ), and inactivated with formaldehyde. Each 0.5 mL dose of vaccine contains
  * NYMC X-179A (A/California/7/2009) (H1N1) - 15μg hemagglutinin (HA)
  * NYMC X-263B (A/HongKong/4801/2014) (H3N2) - 15μg HA
  * NYMC BX-35 (B/Brisbane/60/2008) (B) - 15μg HA
  Arms: Vaccine
Other: Placebo — Phosphate buffered saline with pH 7.2; 0.5 ml/per dose
  Arms: Placebo

SUMMARY:
This Phase 2/3 study assessed whether a single dose of seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) is safe and well-tolerated in adults 18 to 60 years of age; and whether it will induce immune responses to each of the 3 vaccine antigens to meet 1 or both age group-specific Vietnam Ministry of Health (MOH) licensure requirements.

DETAILED DESCRIPTION:
Seasonal influenza viruses circulate widely and cause disease in humans every year. Seasonal influenza viruses evolve continuously, which means that people can get infected multiple times throughout their lives. Therefore the components of seasonal influenza vaccines are reviewed frequently (currently biannually) and updated periodically to ensure continued effectiveness of the vaccines. The World Health Organization (WHO) recommended that influenza vaccines for use in the 2016-2017 northern hemisphere influenza season contain the following viruses:

* NYMC BX-35 reassortant of B/Brisbane/60/2008 (B)
* NYMC X-179A reassortant of A/California/7/2009 (H1N1)
* NYMC X-263B reassortant of H3/A/Hong Kong/4801/2014 (H3N2)

Among circulating influenza B viruses, there were 2 distinct lineages. The B/Brisbane/60/2008-like viruses were from the influenza B/Victoria lineage and represented the predominant circulating influenza B virus. The preclinical evaluation was conducted with all 3 lots of seasonal vaccine used in the Phase 1 study.The Phase 1 study of the IVACFLU-S that was completed in March 2016 identified no safety concerns and demonstrated the vaccine to be highly immunogenic. Given the promising findings, the current study proposed to expand on the safety data of the vaccine, to confirm the immunological findings, and by including individuals up to age 60 to seek regulatory approval for indication in nonelderly adults based on the Vietnam MOH Guidance on Clinical Trial of Influenza Vaccine serological criteria for assessing seasonal influenza.

Phase 2 was conducted at 1 site (District Health Center of Ben Luc, Long An, Vietnam). Subjects were from two age groups: 18-45 years and 46-60 years. Vaccine safety was determined by the Protocol Safety Review Team (PSRT) and approved by Vietnam Ministry of Health (MOH) before starting Phase 3.

Phase 3 was conducted at 2 sites: District Health Center (DHC) of Ben Luc, Long An, Vietnam; and DHC of Long Thanh, Dong Nai. Subjects were from two age groups: 18-45 years and 46-60 years. Both safety and immunogenicity were assessed.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 through 60 years on the day of screening/enrollment.
* Literate (by self-report) and willing to provide written informed consent.
* Able to attend all scheduled visits and to comply with all study procedures.
* Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable under controlled or unchanged for the past 3 months. If medication is used to treat the condition, the medication dose must have been stable for at least 1 month preceding vaccination.

For female subjects:

* Not breastfeeding or pregnant (based on negative urine pregnancy test) or plan to become pregnant up to Day 22. Women who are not surgically sterile (hysterectomy or tubal ligation) or post-menopausal for more than 1 year must have negative pregnancy test and, be willing to utilize reliable birth control measures (intrauterine device, hormonal contraception, condom or diaphragm with spermicide) through the Day 22 visit.

Exclusion criteria:

* Current or recent (within 2 weeks of enrollment) acute severe illness with or without fever.
* Participation in another clinical study involving any therapy within the previous 3 months or planned enrollment in such a study during the period of this study.
* Receipt of any non-study vaccine within 4 weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 22 visit.
* Received seasonal influenza vaccine in last 6 months
* Receipt of immune globulin or other blood products within 3 months prior to study enrollment or planned receipt of such products prior to the Day 22 visit.
* Known or suspected congenital or acquired immunodeficiency.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within 6 months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, ≥ 0.5 mg/kg/day; topical steroids are allowed).
* Unstable illness by history or physical examination that in the opinion of the Investigator, might interfere with the conduct or results of the study or pose additional risk to the subject.
* Hypersensitivity after previous administration of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein, and rubber (from the vaccine vial stoppers).
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion.
* Known active tuberculosis or symptoms of active tuberculosis, regardless of cause (self-report).
* Current alcohol or drug addiction that in the opinion of the Investigator, might interfere with the ability to comply with study procedures.
* History of Guillain-Barré Syndrome
* Neoplastic disease or any hematologic malignancy.
* Any condition that, in the opinion of the Investigator, would increase the health risk to the subject if he/she participates in the study, or would interfere with the evaluation of the study objectives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 889 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phan Cong Hung, MD, Principal Investigator — Pasteur Institute, Ho Chi Minh City
Locations (1):
- Pasteur Institute, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lan PT, Toan NT, Thang HA, Thang TC, Be LV, Thai DH, Huong VM, Nga NT, Tang Y, Holt R, Francesco BS, Flores J, Tewari T. A phase 2/3 double-blind, randomized, placebo-controlled study to evaluate the safety and immunogenicity of a seasonal trivalent inactivated split-virion influenza vaccine (IVACFLU-S) in healthy adults in Vietnam. Hum Vaccin Immunother. 2019;15(12):2933-2939. doi: 10.1080/21645515.2019.1613127. Epub 2019 Jun 20. PMID 31070986

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 2 was conducted at the District Health Center (DHC) of Ben Luc, Long An Province and involved 252 subjects. After positive safety review of Day 8 data, Phase 3 was at 2 sites: the DHC of Ben Luc, Long An Province and the DHC of Long Thanh, Dong Nai Province.
  In total, of the 1399 subjects who were screened, 888 subjects were rand
Groups:
- Vaccine: IVACFLU-S: Trivalent inactivated split virion influenza vaccine
- Placebo: PBS with pH 7.2; 0.5 ml/per dose
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started | 741 | 148
Withdrawal Before Vaccination (Voluntary withdrawal.) | 1 | 0
Vaccinated | 740 | 148
Completed | 738 | 148
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal prior to vaccination | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 740 | 148 | 888
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [18 to 60] | 42.8 [18 to 60] | 42.8 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 431 | 89 | 520
  Male | 309 | 59 | 368
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Kinh | 735 | 148 | 883
  Khmer | 0 | 0 | 0
  Hoa | 2 | 0 | 2
  Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Vietnam | 740 | 148 | 888

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects Experiencing Solicited Local Adverse Events (AE)
Description: Solicited local AEs were assessed by study staff 30 minutes after vaccination.
Time Frame: Within 30 minutes of vaccination
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  Induration | 1 | 0
  Redness | 1 | 0
  Pain | 24 | 0
  Swelling | 1 | 0
  Tenderness | 14 | 1
  No report of solicited local AE | 711 | 147

2. Primary Outcome: Number and Percentage of Subjects Experiencing Solicited Systemic Adverse Events (AE)
Description: Solicited systemic AEs were assessed by study staff 30 minutes after vaccination.
Time Frame: Within 30 minutes of vaccination
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  Chills | 0 | 0
  Fatigue/Malaise | 0 | 0
  Generalized muscle aches | 5 | 0
  Headaches | 1 | 0
  Joint aches | 0 | 0
  Nausea | 1 | 0
  Vomiting | 0 | 0
  No report of solicited systemic AEs | 733 | 148

3. Primary Outcome: Number and Percentage of Subjects Experiencing Solicited Local Adverse Events (AE), by Severity
Description: Solicited local AEs were assessed by study staff 30 minutes after vaccination then daily for 7 days by the subjects. Subjects were provided a thermometer, ruler and a diary to record the presence or absence of solicited AEs, severity of the solicited AE and use of concomitant medication. AEs were graded as follows:
  * Mild: Mild symptoms causing no or minimal interference with usual social and functional activities with intervention not indicated.
  * Moderate: Moderate symptoms causing greater than minimal interference with usual social and functional activities with intervention indicated.
  * Severe: Severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated.
  * Life-threatening: Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: Day 1 to Day 7
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  Hardness: Mild | 23 | 0
  Hardness: Moderate | 1 | 0
  Hardness: Severe | 0 | 0
  Hardness: Life threatening | 0 | 0
  Hardness: None reported | 716 | 148
  Pain: Mild | 405 | 25
  Pain: Moderate | 55 | 1
  Pain: Severe | 1 | 0
  Pain: Life threatening | 0 | 0
  Pain: None reported | 279 | 122
  Redness: Mild | 18 | 1
  Redness: Moderate | 1 | 0
  Redness: Severe | 0 | 0
  Redness: Life threatening | 0 | 0
  Redness: None reported | 721 | 147
  Swelling: Mild | 20 | 1
  Swelling: Moderate | 6 | 0
  Swelling: Severe | 0 | 0
  Swelling: Life threatening | 0 | 0
  Swelling: None reported | 714 | 147
  Tenderness: Mild | 441 | 30
  Tenderness: Moderate | 54 | 2
  Tenderness: Severe | 1 | 0
  Tenderness: Life threatening | 0 | 0
  Tenderness: None reported | 244 | 116

4. Primary Outcome: Number and Percentage of Subjects Experiencing Solicited Systemic Adverse Events (AE), by Severity
Description: Solicited systemic AEs were assessed by study staff 30 minutes after vaccination then daily for 7 days by the subjects. Subjects were provided a thermometer, ruler and a diary to record the presence or absence of solicited AEs, severity of the solicited AE and use of concomitant medication. AEs were graded as follows:
  * Mild: Mild symptoms causing no or minimal interference with usual social and functional activities with intervention not indicated.
  * Moderate: Moderate symptoms causing greater than minimal interference with usual social and functional activities with intervention indicated.
  * Severe: Severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated.
  * Life-threatening: Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: Day 1 to Day 7
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  Chills: Mild | 36 | 10
  Chills: Moderate | 9 | 2
  Chills: Severe | 0 | 1
  Chills: Life threatening | 0 | 0
  Chills: None reported | 695 | 135
  Fatigue/Malaise: Mild | 111 | 18
  Fatigue/Malaise: Moderate | 29 | 8
  Fatigue/Malaise: Severe | 2 | 1
  Fatigue/Malaise: Life threatening | 0 | 0
  Fatigue/Malaise: None reported | 598 | 121
  Generalized muscle aches: Mild | 114 | 14
  Generalized muscle aches: Moderate | 23 | 1
  Generalized muscle aches: Severe | 0 | 1
  Generalized muscle aches: Life threatening | 0 | 0
  Generalized muscle aches: None reported | 603 | 132
  Headaches: Mild | 93 | 23
  Headaches: Moderate | 27 | 4
  Headaches: Severe | 1 | 2
  Headaches: Life threatening | 0 | 0
  Headaches: None reported | 619 | 119
  Joint aches: Mild | 42 | 11
  Joint aches: Moderate | 16 | 0
  Joint aches: Severe | 0 | 1
  Joint aches: Life threatening | 0 | 0
  Joint aches: None reported | 682 | 136
  Nausea: Mild | 14 | 4
  Nausea: Moderate | 2 | 0
  Nausea: Severe | 1 | 1
  Nausea: Life threatening | 0 | 0
  Nausea: None reported | 723 | 143
  Vomiting: Mild | 3 | 0
  Vomiting: Moderate | 2 | 0
  Vomiting: Severe | 1 | 0
  Vomiting: Life threatening | 0 | 0
  Vomiting: None reported | 734 | 148

5. Primary Outcome: Number and Percentage of Subjects Experiencing Fever
Description: Subjects reporting body temperature by maximum severity; Grade 0: <38°C, Grade 1: 38.0 - <38.6°C, Grade 2: 38.6 - <39.3°C, Grade 3: 39.3 - <40.0°C, Grade 4: >= 40.0°C
Time Frame: Day 1 to Day 7
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  Grade 0 | 729 | 146
  Grade 1 | 5 | 1
  Grade 2 | 5 | 1
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0

6. Primary Outcome: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events (AE)
Description: Unsolicited AEs were observed by study staff while the subject is at a clinic for a study visit or reported by the subject at any time. Any sign or symptom that would normally be considered a "solicited AE" (for example, fever, nausea, injection site pain) starting after 7 days post-vaccination was to be recorded as an unsolicited AE. The clinician determined whether there was a reasonable possibility that the investigational product(s) caused or contributed to an AE. The following guidelines were used:
  * Related: There is a reasonable possibility that the study vaccine caused the AE. "Reasonable possibility" means that there is evidence to suggest a causal relationship between the study product and the AE.
  * Not Related: There is not a reasonable possibility that the administration of the study product caused the event.
Time Frame: Day 1 to Day 21
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  At least one unsolicited AE | 110 | 17
  At least one vaccine-related unsolicited AE | 3 | 1
  At least one severe unsolicited AE | 2 | 0
  At least one life threatening unsolicited AE | 0 | 0
  Subjects requiring treatment during the study | 64 | 11

7. Primary Outcome: Number and Percentage of Subjects Experiencing Unsolicited Serious Adverse Events (SAE)
Description: as for outcome 6
Time Frame: Day 1 to Day 91
Population: All recipients of the vaccine in Phases 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 740 | 148
Participants
  Related to vaccine | 0 | 0
  Not related to vaccine | 4 | 2

8. Primary Outcome: Number and Percentage of Subjects With Seroconversion of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens, Overall and by Age Group
Description: Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine (A/H1N1, B, and A/H3N2). This testing was performed by VisMederi SRL laboratory (Siena, Italy), by using a validated assay. Sample collection on Day 1 was prior to administration of study product.
  Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:
  * pre-vaccination titer < 1:10 and a post-vaccination titer measured on Day 22 of ≥ 1:40, or
  * pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination measured on Day 22
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were participated in the study through at least day 22, overall and by age group.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 209 | 42
Participants
  Overall: A/H1N1 | 147 | 0
  Overall: A/H3N2 | 159 | 0
  Overall: B | 113 | 1
  Ages 18-45: A/H1N1: number analyzed (Participants) | 104 | 21
  Ages 18-45: A/H1N1 | 73 | 0
  Ages 18-45: AH3N2: number analyzed (Participants) | 104 | 21
  Ages 18-45: AH3N2 | 74 | 0
  Ages 18-45: B: number analyzed (Participants) | 104 | 21
  Ages 18-45: B | 52 | 0
  Ages 46-60: A/H1N1: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H1N1 | 74 | 0
  Ages 46-60: A/H3N2: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H3N2 | 85 | 0
  Ages 46-60: B: number analyzed (Participants) | 105 | 21
  Ages 46-60: B | 61 | 1

9. Primary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens at Baseline and Day 22, Overall and by Age Group
Description: Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine (A/H1N1, B, and A/H3N2). This testing was performed by VisMederi SRL laboratory (Siena, Italy), by using a validated assay. Sample collection on Day 1 was prior to administration of study product.
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were participated in the study through at least day 22, overall and by age group.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 209 | 42
titer
  Overall: A/H1N1: Day 1 | 9.93 [8.593 to 11.465] | 13.51 [9.288 to 19.665]
  Overall: A/H1N1: Day 22 | 130.48 [107.898 to 157.78] | 13.46 [9.438 to 19.192]
  Overall: A/H3N2: Day 1 | 12.92 [11.256 to 14.831] | 12.65 [8.836 to 18.115]
  Overall: A/H3N2: Day 22 | 153.12 [127.996 to 183.17] | 12.65 [8.859 to 18.068]
  Overall: B: Day 1 | 7.17 [6.620 to 7.756] | 6.35 [5.468 to 7.379]
  Overall: B: Day 22 | 42.04 [35.654 to 49.570] | 6.79 [5.580 to 8.251]
  Ages 18-45: A/H1N1: Day 1: number analyzed (Participants) | 104 | 21
  Ages 18-45: A/H1N1: Day 1 | 12.65 [10.102 to 15.837] | 15.49 [8.399 to 28.553]
  Ages 18-45: A/H1N1: Day 22: number analyzed (Participants) | 104 | 21
  Ages 18-45: A/H1N1: Day 22 | 149.19 [119.134 to 186.81] | 15.74 [8.732 to 28.386]
  Ages 18-45: A/H3N2: Day 1: number analyzed (Participants) | 104 | 21
  Ages 18-45: A/H3N2: Day 1 | 16.16 [13.008 to 20.072] | 21.36 [11.900 to 38.359]
  Ages 18-45: A/H3N2: Day 22: number analyzed (Participants) | 104 | 21
  Ages 18-45: A/H3N2: Day 22 | 145.26 [114.633 to 184.07] | 22.26 [12.528 to 39.569]
  Ages 18-45: B: Day 1: number analyzed (Participants) | 104 | 21
  Ages 18-45: B: Day 1 | 6.48 [5.915 to 7.108] | 6.20 [5.273 to 7.282]
  Ages 18-45: B: Day 22: number analyzed (Participants) | 104 | 21
  Ages 18-45: B: Day 22 | 38.18 [30.703 to 47.469] | 6.62 [5.278 to 8.302]
  Ages 46-60: A/H1N1: Day 1: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H1N1: Day 1 | 7.81 [6.569 to 9.278] | 11.79 [7.278 to 19.112]
  Ages 46-60: A/H1N1: Day 22: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H1N1: Day 22 | 114.26 [84.025 to 155.382] | 11.51 [7.418 to 17.846]
  Ages 46-60: A/H3N2: Day 1: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H3N2: Day 1 | 10.35 [8.790 to 12.193] | 7.49 [5.447 to 10.304]
  Ages 46-60: A/H3N2: Day 22: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H3N2: Day 22 | 161.33 [122.860 to 211.83] | 7.19 [5.363 to 9.635]
  Ages 46-60: B: Day 1: number analyzed (Participants) | 105 | 21
  Ages 46-60: B: Day 1 | 7.91 [6.964 to 8.986] | 6.51 [4.979 to 8.514]
  Ages 46-60: B: Day 22: number analyzed (Participants) | 105 | 21
  Ages 46-60: B: Day 22 | 46.25 [36.051 to 59.341] | 6.96 [4.950 to 9.773]

10. Primary Outcome: Geometric Mean Fold Change of Serum Hemagglutination Inhibition (HAI) Antibody Titer, Overall and by Age Group
Description: Fold change in titer between Day 1 and Day 22. Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine (A/H1N1, B, and A/H3N2). This testing was performed by VisMederi SRL laboratory (Siena, Italy), by using a validated assay. Sample collection on Day 1 was prior to administration of study product.
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were participated in the study through at least day 22, overall and by age group.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 209 | 42
fold change
  Overall: A/H1N1 | 13.15 [10.623 to 16.268] | 1.00 [0.909 to 1.091]
  Overall: A/H3N2 | 11.85 [9.762 to 14.388] | 1.00 [0.939 to 1.065]
  Overall: B | 5.87 [4.987 to 6.902] | 1.07 [0.895 to 1.275]
  Ages 18-45: A/H1N1: number analyzed (Participants) | 104 | 21
  Ages 18-45: A/H1N1 | 11.79 [8.832 to 15.752] | 1.02 [0.852 to 1.213]
  Ages 18-45: AH3N2: number analyzed (Participants) | 104 | 21
  Ages 18-45: AH3N2 | 8.99 [6.878 to 11.750] | 1.04 [0.935 to 1.162]
  Ages 18-45: B: number analyzed (Participants) | 104 | 21
  Ages 18-45: B | 5.89 [4.694 to 7.385] | 1.07 [0.852 to 1.340]
  Ages 46-60: A/H1N1: number analyzed (Participants) | 105 | 21
  Ages 46-60: A/H1N1 | 14.64 [10.669 to 20.078] | 0.98 [0.908 to 1.048]
  Ages 46-60: AH3N2: number analyzed (Participants) | 105 | 21
  Ages 46-60: AH3N2 | 15.58 [11.839 to 20.512] | 0.96 [0.895 to 1.029]
  Ages 46-60: B: number analyzed (Participants) | 105 | 21
  Ages 46-60: B | 5.85 [4.615 to 7.407] | 1.07 [0.797 to 1.433]

11. Secondary Outcome: Number and Percentage of Subjects With at Least a 4-fold Increase in HAI Antibody Titer, by Strain, Age Group, and Baseline Titer
Description: as for outcome 9
Time Frame: Day 22
Population: Phase 3 participants who were participated in the study through at least day 22, overall and by age group.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 209 | 42
Participants
  Overall A/H1N1; baseline <1:10: number analyzed (Participants) | 131 | 20
  Overall A/H1N1; baseline <1:10 | 97 | 0
  Overall for A/H1N1; baseline ≥1:10: number analyzed (Participants) | 78 | 22
  Overall for A/H1N1; baseline ≥1:10 | 50 | 0
  Overall A/H3N2; baseline <1:10: number analyzed (Participants) | 90 | 21
  Overall A/H3N2; baseline <1:10 | 66 | 0
  Overall A/H3N2; baseline ≥1:10: number analyzed (Participants) | 119 | 21
  Overall A/H3N2; baseline ≥1:10 | 93 | 0
  Overall B; baseline <1:10: number analyzed (Participants) | 139 | 32
  Overall B; baseline <1:10 | 71 | 1
  Overall B; baseline ≥1:10: number analyzed (Participants) | 70 | 10
  Overall B; baseline ≥1:10 | 42 | 0
  Age18-45 A/H1N1; baseline <1:10: number analyzed (Participants) | 55 | 10
  Age18-45 A/H1N1; baseline <1:10 | 45 | 0
  Age 18-45 A/H1N1; baseline ≥1:10: number analyzed (Participants) | 49 | 11
  Age 18-45 A/H1N1; baseline ≥1:10 | 28 | 0
  Age18-45 A/H3N2; baseline <1:10: number analyzed (Participants) | 36 | 6
  Age18-45 A/H3N2; baseline <1:10 | 26 | 0
  Age 18-45 A/H3N2; baseline ≥1:10: number analyzed (Participants) | 68 | 15
  Age 18-45 A/H3N2; baseline ≥1:10 | 48 | 0
  Age18-45 B; baseline <1:10: number analyzed (Participants) | 76 | 15
  Age18-45 B; baseline <1:10 | 38 | 0
  Age 18-45 B; baseline ≥1:10: number analyzed (Participants) | 28 | 6
  Age 18-45 B; baseline ≥1:10 | 14 | 0
  Age 46-60 A/H1N1; baseline <1:10: number analyzed (Participants) | 76 | 10
  Age 46-60 A/H1N1; baseline <1:10 | 52 | 0
  Age 46-60 A/H1N1; baseline ≥1:10: number analyzed (Participants) | 29 | 11
  Age 46-60 A/H1N1; baseline ≥1:10 | 22 | 0
  Age 46-60 A/H3N2; baseline <1:10: number analyzed (Participants) | 54 | 15
  Age 46-60 A/H3N2; baseline <1:10 | 40 | 0
  Age 46-60 A/H3N2; baseline ≥1:10: number analyzed (Participants) | 51 | 6
  Age 46-60 A/H3N2; baseline ≥1:10 | 45 | 0
  Age 46-60 B; baseline <1:10: number analyzed (Participants) | 63 | 17
  Age 46-60 B; baseline <1:10 | 33 | 1
  Age 46-60 B; baseline ≥1:10: number analyzed (Participants) | 42 | 4
  Age 46-60 B; baseline ≥1:10 | 28 | 0

12. Secondary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens at Baseline and Day 22: All Subjects
Description: Serum specimens during Phase 3 were tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine (A/H1N1, B, and A/H1N1). This testing was performed by VisMederi SRL laboratory (Siena, Italy), by using a validated assay. Sample collection on Day 1 was prior to administration of study product.
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were participated in the study through at least day 22.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 209 | 42
titer
  A/H1N1, Day 1: baseline <1:10: number analyzed (Participants) | 131 | 20
  A/H1N1, Day 1: baseline <1:10 | 5 (1) | 5 (1)
  A/H1N1, Day 1: baseline ≥1:10: number analyzed (Participants) | 78 | 22
  A/H1N1, Day 1: baseline ≥1:10 | 31.40 (2.55) | 33.37 (2.76)
  A/H1N1, Day 22: baseline <1:10: number analyzed (Participants) | 131 | 20
  A/H1N1, Day 22: baseline <1:10 | 99.78 (4.88) | 5.45 (1.31)
  A/H1N1, Day 22: baseline ≥1:10: number analyzed (Participants) | 78 | 22
  A/H1N1, Day 22: baseline ≥1:10 | 204.75 (2.27) | 30.60 (2.69)
  A/H3N2 Day 1: baseline <1:10: number analyzed (Participants) | 90 | 21
  A/H3N2 Day 1: baseline <1:10 | 5 (1) | 5 (1)
  A/H3N2 Day 1: baseline ≥1:10: number analyzed (Participants) | 119 | 21
  A/H3N2 Day 1: baseline ≥1:10 | 26.49 (2.16) | 32.01 (2.60)
  A/H3N2 Day 22: baseline <1:10: number analyzed (Participants) | 90 | 21
  A/H3N2 Day 22: baseline <1:10 | 97.17 (4.72) | 5 (1)
  A/H3N2 Day 22: baseline ≥1:10: number analyzed (Participants) | 119 | 21
  A/H3N2 Day 22: baseline ≥1:10 | 215.97 (2.65) | 32.01 (2.54)
  B, Day 1: baseline <1:10: number analyzed (Participants) | 139 | 32
  B, Day 1: baseline <1:10 | 5 (1) | 5 (1)
  B, Day 1: baseline ≥1:10: number analyzed (Participants) | 70 | 10
  B, Day 1: baseline ≥1:10 | 14.64 (1.63) | 13.66 (1.56)
  B, Day 22: baseline <1:10: number analyzed (Participants) | 139 | 32
  B, Day 22: baseline <1:10 | 33.10 (3.45) | 5.95 (1.80)
  B, Day 22: baseline ≥1:10: number analyzed (Participants) | 70 | 10
  B, Day 22: baseline ≥1:10 | 67.61 (2.71) | 10.35 (1.78)

13. Secondary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens at Baseline and Day 22: Subjects Aged 18-45
Description: as for outcome 9
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were age 18-45 and participated in the study through at least day 22.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 104 | 21
titer
  A/H1N1, Day 1: baseline <1:10: number analyzed (Participants) | 55 | 10
  A/H1N1, Day 1: baseline <1:10 | 5 (1) | 5 (1)
  A/H1N1, Day 1: baseline ≥1:10: number analyzed (Participants) | 49 | 11
  A/H1N1, Day 1: baseline ≥1:10 | 35.85 (2.41) | 43.28 (2.95)
  A/H1N1, Day 22: baseline <1:10: number analyzed (Participants) | 55 | 10
  A/H1N1, Day 22: baseline <1:10 | 117.13 (4.11) | 5.95 (1.45)
  A/H1N1, Day 22: baseline ≥1:10: number analyzed (Participants) | 49 | 11
  A/H1N1, Day 22: baseline ≥1:10 | 195.73 (2) | 38.15 (3.29)
  A/H3N2 Day 1: baseline <1:10: number analyzed (Participants) | 36 | 6
  A/H3N2 Day 1: baseline <1:10 | 5 (1) | 5 (1)
  A/H3N2 Day 1: baseline ≥1:10: number analyzed (Participants) | 68 | 15
  A/H3N2 Day 1: baseline ≥1:10 | 30.07 (2.42) | 38.19 (2.85)
  A/H3N2 Day 22: baseline <1:10: number analyzed (Participants) | 36 | 6
  A/H3N2 Day 22: baseline <1:10 | 88.51 (4.49) | 5 (1)
  A/H3N2 Day 22: baseline ≥1:10: number analyzed (Participants) | 68 | 15
  A/H3N2 Day 22: baseline ≥1:10 | 188.82 (2.58) | 40.46 (2.64)
  B, Day 1: baseline <1:10: number analyzed (Participants) | 76 | 15
  B, Day 1: baseline <1:10 | 5 (1) | 5 (1)
  B, Day 1: baseline ≥1:10: number analyzed (Participants) | 28 | 6
  B, Day 1: baseline ≥1:10 | 13.13 (1.46) | 10.59 (1.15)
  B, Day 22: baseline <1:10: number analyzed (Participants) | 76 | 15
  B, Day 22: baseline <1:10 | 34.97 (3.22) | 6.02 (1.66)
  B, Day 22: baseline ≥1:10: number analyzed (Participants) | 28 | 6
  B, Day 22: baseline ≥1:10 | 48.46 (2.59) | 8.41 (1.53)

14. Secondary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) Antibodies for Vaccine Antigens at Baseline and Day 22: Subjects Aged 46-60
Description: as for outcome 9
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were age 46-60 and participated in the study through at least day 22.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 105 | 21
titer
  A/H1N1, Day 1: baseline <1:10: number analyzed (Participants) | 76 | 10
  A/H1N1, Day 1: baseline <1:10 | 5 (1) | 5 (1)
  A/H1N1, Day 1: baseline ≥1:10: number analyzed (Participants) | 29 | 11
  A/H1N1, Day 1: baseline ≥1:10 | 25.10 (2.72) | 25.73 (2.50)
  A/H1N1, Day 22: baseline <1:10: number analyzed (Participants) | 76 | 10
  A/H1N1, Day 22: baseline <1:10 | 88.85 (5.47) | 5 (1)
  A/H1N1, Day 22: baseline ≥1:10: number analyzed (Participants) | 29 | 11
  A/H1N1, Day 22: baseline ≥1:10 | 220.93 (2.74) | 24.55 (2.08)
  A/H3N2 Day 1: baseline <1:10: number analyzed (Participants) | 54 | 15
  A/H3N2 Day 1: baseline <1:10 | 5 (1) | 5 (1)
  A/H3N2 Day 1: baseline ≥1:10: number analyzed (Participants) | 51 | 6
  A/H3N2 Day 1: baseline ≥1:10 | 22.37 (1.74) | 20.59 (1.64)
  A/H3N2 Day 22: baseline <1:10: number analyzed (Participants) | 54 | 15
  A/H3N2 Day 22: baseline <1:10 | 103.41 (4.93) | 5 (1)
  A/H3N2 Day 22: baseline ≥1:10: number analyzed (Participants) | 51 | 6
  A/H3N2 Day 22: baseline ≥1:10 | 258.34 (2.70) | 17.82 (1.69)
  B, Day 1: baseline <1:10: number analyzed (Participants) | 63 | 17
  B, Day 1: baseline <1:10 | 5 (1) | 5 (1)
  B, Day 1: baseline ≥1:10: number analyzed (Participants) | 42 | 4
  B, Day 1: baseline ≥1:10 | 15.74 (1.72) | 20 (1.63)
  B, Day 22: baseline <1:10: number analyzed (Participants) | 63 | 17
  B, Day 22: baseline <1:10 | 30.97 (3.75) | 5.89 (1.96)
  B, Day 22: baseline ≥1:10: number analyzed (Participants) | 42 | 4
  B, Day 22: baseline ≥1:10 | 84.41 (2.64) | 14.14 (2)

15. Secondary Outcome: Geometric Mean Fold Change in HAI Antibody Titer, by Strain, Age Group, and Baseline Titer
Description: as for outcome 9
Time Frame: Day 1, Day 22
Population: Phase 3 participants who were participated in the study through at least day 22, overall and by age group.
Measure: Geometric Mean (Standard Deviation); unit: fold change
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 209 | 42
fold change
  Overall A/H1N1; baseline <1:10: number analyzed (Participants) | 131 | 20
  Overall A/H1N1; baseline <1:10 | 19.96 (4.88) | 1.09 (1.31)
  Overall for A/H1N1; baseline ≥1:10: number analyzed (Participants) | 78 | 22
  Overall for A/H1N1; baseline ≥1:10 | 6.52 (3.48) | 0.92 (1.34)
  Overall A/H3N2; baseline <1:10: number analyzed (Participants) | 90 | 21
  Overall A/H3N2; baseline <1:10 | 19.43 (4.72) | 1 (1)
  Overall A/H3N2; baseline ≥1:10: number analyzed (Participants) | 119 | 21
  Overall A/H3N2; baseline ≥1:10 | 8.15 (3.30) | 1 (1)
  Overall B; baseline <1:10: number analyzed (Participants) | 139 | 32
  Overall B; baseline <1:10 | 6.62 (3.45) | 1.19 (1.80)
  Overall B; baseline ≥1:10: number analyzed (Participants) | 70 | 10
  Overall B; baseline ≥1:10 | 4.62 (2.89) | 0.76 (1.38)
  Age18-45 A/H1N1; baseline <1:10: number analyzed (Participants) | 55 | 10
  Age18-45 A/H1N1; baseline <1:10 | 23.43 (4.11) | 1.19 (1.45)
  Age 18-45 A/H1N1; baseline ≥1:10: number analyzed (Participants) | 49 | 11
  Age 18-45 A/H1N1; baseline ≥1:10 | 5.46 (3.20) | 0.88 (1.43)
  Age18-45 A/H3N2; baseline <1:10: number analyzed (Participants) | 36 | 6
  Age18-45 A/H3N2; baseline <1:10 | 17.70 (4.49) | 1.00 (1.00)
  Age 18-45 A/H3N2; baseline ≥1:10: number analyzed (Participants) | 68 | 15
  Age 18-45 A/H3N2; baseline ≥1:10 | 6.28 (3.21) | 1.06 (1.33)
  Age18-45 B; baseline <1:10: number analyzed (Participants) | 76 | 15
  Age18-45 B; baseline <1:10 | 6.99 (3.22) | 1.20 (1.66)
  Age 18-45 B; baseline ≥1:10: number analyzed (Participants) | 28 | 6
  Age 18-45 B; baseline ≥1:10 | 3.69 (2.81) | 0.79 (1.43)
  Age 46-60 A/H1N1; baseline <1:10: number analyzed (Participants) | 76 | 10
  Age 46-60 A/H1N1; baseline <1:10 | 17.77 (5.47) | 1.00 (1.00)
  Age 46-60 A/H1N1; baseline ≥1:10: number analyzed (Participants) | 29 | 11
  Age 46-60 A/H1N1; baseline ≥1:10 | 8.80 (3.84) | 0.95 (1.25)
  Age 46-60 A/H3N2; baseline <1:10: number analyzed (Participants) | 54 | 15
  Age 46-60 A/H3N2; baseline <1:10 | 20.68 (4.93) | 1.00 (1.00)
  Age 46-60 A/H3N2; baseline ≥1:10: number analyzed (Participants) | 51 | 6
  Age 46-60 A/H3N2; baseline ≥1:10 | 11.55 (3.16) | 0.87 (1.32)
  Age 46-60 B; baseline <1:10: number analyzed (Participants) | 63 | 17
  Age 46-60 B; baseline <1:10 | 6.19 (3.75) | 1.18 (1.96)
  Age 46-60 B; baseline ≥1:10: number analyzed (Participants) | 42 | 4
  Age 46-60 B; baseline ≥1:10 | 5.36 (2.90) | 0.71 (1.33)

ADVERSE EVENTS:
Time Frame: 22 days for non-serious adverse events; 91 days for serious adverse events.
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/740 | 0/148
Serious Adverse Events (participants affected / at risk) | 4/740 | 2/148
Other Adverse Events (participants affected / at risk) | 110/740 | 17/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=740) | Placebo (N=148)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=740) | Placebo (N=148)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gingival Swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection Site Haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection Site Pruritus (General disorders) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Food Allergy (Immune system disorders) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 8 (8) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Intercostal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 11 (11) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03095599/Prot_SAP_ICF_000.pdf